CLINICAL TRIAL: NCT02441998
Title: Prospective Multi-Center Study Evaluating Real-Time Characterizations of Diminutive Colorectal Polyps Using Narrow Band Imaging: Implications for the Resect and Discard Strategy
Brief Title: Real-Time Characterizations of Diminutive Colorectal Polyps Using Narrow Band Imaging
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Swati Patel, Clinical Lecturer, University of Michigan
Other Study IDs: 131998
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Diminutive Polyps; Narrow Band Imaging; Colonic Polyps; colonoscopy; diagnostic imaging; optical diagnosis
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Education intervention: Training in Narrow Band Imaging — Two hour training session in interpretation and application of narrow band imaging technology

SUMMARY:
Colorectal cancer is the second leading cause of cancer related death in the United States. Colonoscopy is the most commonly performed screening procedure and diminutive polyps (<5mm) are the most commonly found polyps during colonoscopy. Although these polyps have a very low risk of harboring malignancy, they are routinely removed to determine surveillance intervals.

Narrow Band Imaging is equipped on widely available colonoscopes and in expert hands can allow accurate real-time optical histologic diagnosis of colorectal polyps. If this practice can be applied widely, there is significant potential for cost savings.

This has led to a 'characterize, resect and discard' strategy where polyps determined to be hyperplastic (benign with no neoplastic potential) can be left in place and those determined to be adenomatous (have neoplastic potential) can be resected and discarded.

It is unclear if endoscopists without prior expertise or training in Narrow Band Imaging can achieve adequate diagnostic accuracy to put 'characterize, resect and discard' into wide practice.

DETAILED DESCRIPTION:
Gastroenterologists without prior training in NBI from two affiliated academic hospitals will participate in an ex-vivo training session in which they will view a short audiovisual tool describing previously validated NBI criteria to determine polyp histology, followed by reviewing 80 videos of diminutive polyps under NBI and will record predicted polyp histology and degree of confidence. After each video, targeted feedback regarding actual polyp histology and NBI criteria supporting the diagnosis will be provided. Participants will then employ NBI in real-time colonoscopy (in-vivo) and record predicted polyp histology, degree of confidence and predicted surveillance intervals based on NBI interpretations. Each study polyp will be sent for histology separately. Performance will be assessed by comparing predicted histology with actual histology. Structured performance feedback will be given to promote practice-based learning, establish a real-time learning curve and determine the number of observations required to achieve competency in-vivo.

The primary aim of this study was to determine whether endoscopists with no prior experience or training in Narrow Band Imaging can achieve the thresholds set forth by the American Society of Gastrointestinal Endoscopy: For diminutive colorectal polyp diagnoses made with 'high-confidence,' a (1) greater than or equal to 90% negative predictive value in the rectosigmoid colon and a (2) greater than or equal to 90% agreement in surveillance intervals predicted by narrow band imaging and those based on the current gold standard of histology.

The secondary outcomes for the in-vivo phase included (1) evaluating overall group performance (accuracy, sensitivity, specificity, predictive values) of optical diagnoses using NBI based on degree of confidence and location within the colon, (2) evaluating individual performance on the ASGE benchmarks, (3) determining predictors of performance, and (4) determining real-time learning effect in the setting of ongoing, structured performance feedback. The secondary outcomes for the ex-vivo (training) phase included (1) evaluating overall performance by degree of confidence, (2) determining predictors of performance during training and (3) evaluating a learning effect in the setting of ongoing feedback during training.

Sample size was calculated to show an NPV of 90% or higher assuming that the true NPV is 95% for rectosigmoid polyps characterized with "high-confidence," based on 26 participating endoscopists and within-endoscopist correlation of 0.05. This will require 336 total rectosigmoid non-adenoma polyps characterized with "high-confidence," and assuming approximately 22% rectosigmoid polyps, 70% with high confidence and 80% hyperplastic, the study will require approximately 2,727 polyps and 1,364 colonoscopies in total, assuming approximately two polyps per colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Active member of division of Gastroenterology
* Performs colonoscopy
* No prior training in Narrow Band Imaging
* Informed consent to participate

Exclusion Criteria:

* Low annual colonoscopy volume (<200 per year)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Practicing gastroenterologists from 2 academic medical centers
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
ASGE PIVI Thresholds: >90% NPV in rectosigmoid, > 90% agreement in surveillance intervals | 1 year

SECONDARY OUTCOMES:
In vivo overall and individual performance assessed by accuracy, sensitivity, specificity, positive predictive value, negative predictive value | 1 year
Ex vivo overall and individual performance assessed by accuracy, sensitivity, specificity, positive predictive value, negative predictive value | 1 year

REFERENCES:
- [Background] Ladabaum U, Fioritto A, Mitani A, Desai M, Kim JP, Rex DK, Imperiale T, Gunaratnam N. Real-time optical biopsy of colon polyps with narrow band imaging in community practice does not yet meet key thresholds for clinical decisions. Gastroenterology. 2013 Jan;144(1):81-91. doi: 10.1053/j.gastro.2012.09.054. Epub 2012 Oct 3. PMID 23041328
- [Background] Patel SG, Rastogi A, Austin G, Hall M, Siller BA, Berman K, Yen R, Bansal A, Ahnen DJ, Wani S. Gastroenterology trainees can easily learn histologic characterization of diminutive colorectal polyps with narrow band imaging. Clin Gastroenterol Hepatol. 2013 Aug;11(8):997-1003.e1. doi: 10.1016/j.cgh.2013.02.020. Epub 2013 Mar 1. PMID 23466714
- [Background] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Background] Rastogi A, Keighley J, Singh V, Callahan P, Bansal A, Wani S, Sharma P. High accuracy of narrow band imaging without magnification for the real-time characterization of polyp histology and its comparison with high-definition white light colonoscopy: a prospective study. Am J Gastroenterol. 2009 Oct;104(10):2422-30. doi: 10.1038/ajg.2009.403. Epub 2009 Jul 7. PMID 19584829
- [Background] Ignjatovic A, East JE, Suzuki N, Vance M, Guenther T, Saunders BP. Optical diagnosis of small colorectal polyps at routine colonoscopy (Detect InSpect ChAracterise Resect and Discard; DISCARD trial): a prospective cohort study. Lancet Oncol. 2009 Dec;10(12):1171-8. doi: 10.1016/S1470-2045(09)70329-8. Epub 2009 Nov 10. PMID 19910250
- [Background] ASGE Technology Committee; Abu Dayyeh BK, Thosani N, Konda V, Wallace MB, Rex DK, Chauhan SS, Hwang JH, Komanduri S, Manfredi M, Maple JT, Murad FM, Siddiqui UD, Banerjee S. ASGE Technology Committee systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2015 Mar;81(3):502.e1-502.e16. doi: 10.1016/j.gie.2014.12.022. Epub 2015 Jan 16. PMID 25597420
- [Derived] Patel SG, Schoenfeld P, Kim HM, Ward EK, Bansal A, Kim Y, Hosford L, Myers A, Foster S, Craft J, Shopinski S, Wilson RH, Ahnen DJ, Rastogi A, Wani S. Real-Time Characterization of Diminutive Colorectal Polyp Histology Using Narrow-Band Imaging: Implications for the Resect and Discard Strategy. Gastroenterology. 2016 Feb;150(2):406-18. doi: 10.1053/j.gastro.2015.10.042. Epub 2015 Oct 30. PMID 26522260